CLINICAL TRIAL: NCT00808509
Title: A Pilot Study of the Feasibility of Discontinuation of Adalimumab in Stable Rheumatoid Arthritis Patients in Clinical Remission (ADMIRE)
Brief Title: A Pilot Study of the Feasibility of Discontinuation of Adalimumab in Stable Rheumatoid Arthritis Patients in Clinical Remission
Acronym: ADMIRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Pharma Consulting Group AB (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: W10-046; 2008-004398-16 (EudraCT Number)
Record Dates: First submitted 2008-12-12; First posted 2008-12-16 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: adalimumab,Remission,drug discontinuation
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab + MTX (Active Comparator): Participants continued treatment with adalimumab 40 mg subcutaneously every other week plus methotrexate (at least 10 mg/week orally or subcutaneously) for 52 weeks. After Week 52 an observational extension period ensued where participants were treated at the discretion of the investigator.
  Interventions: Biological: adalimumab; Drug: methotrexate
- Methotrexate (Experimental): Participants discontinued adalimumab and continued to receive methotrexate (at least 10 mg/week orally or subcutaneously) for 52 weeks. Participants with a significant increase in RA disease activity were re-instituted to adalimumab 40 mg every other week (rescue arm). After Week 52 an observational extension period ensued where participants were treated at the discretion of the investigator.
  Interventions: Drug: methotrexate

INTERVENTIONS:
Biological: adalimumab — 40 mg every other week via subcutaneous injection
  Other Names: ABT-D2E7; HUMIRA
  Arms: Adalimumab + MTX
Drug: methotrexate — At least 10 mg/week administered orally or subcutaneously

SUMMARY:
The purpose of this pilot study is to investigate the possibility of discontinuing adalimumab therapy in patients with rheumatoid arthritis who are in stable remission after treatment with adalimumab in combination with methotrexate.

DETAILED DESCRIPTION:
Treatments with adalimumab and other tumor necrosis factor (TNF) blockers, once started as therapy for rheumatoid arthritis (RA), are usually continued indefinitely. Information concerning the possibility of discontinuing anti-TNF therapy in RA patients who are in remission is limited. This is a pilot study in one country to study the effect of adalimumab discontinuation. The objective is to assess the proportion of patients with established RA in stable remission (Disease Activity Score [DAS]28 <2.6) after treatment with adalimumab in combination with methotrexate, in whom it is possible to discontinue adalimumab and to compare the remission rates among patients on sustained therapy with adalimumab + methotrexate with remission rates among patients who discontinued adalimumab.

Rheumatoid arthritis patients in stable remission (DAS28 < 2.6) treated with adalimumab + methotrexate were randomized in a 1:1 ratio to continue with adalimumab treatment or discontinue adalimumab treatment for the following 52 weeks. Subsequently an observational extension was conducted to observe patients treated at the discretion of the investigator. The observational extension period lasted until Weeks 105 - 156 (average Week 125) and consisted of one follow-up visit. Participants randomized to discontinue adalimumab therapy will be reinstituted to adalimumab if DAS28-score increases by >1.2 units from baseline and/or is scored ≥2.6 at any visit during the study and will be followed for an additional 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Diagnosis of RA as defined by the 1987-revised American College of Rheumatology (ACR)-classification and has positive rheumatoid factor (RF) test or erosion on X-ray of hands or feet.
* Currently treated with adalimumab and MTX (at least 10 mg/week; orally or subcutaneously).
* In remission as defined by disease activity score (DAS)28 <2.6 for at least the past 3 months.
* Concomitant disease-modifying anti-rheumatic drug (DMARD) or oral corticosteroid therapy has been stable for at least 3 months at study entry.
* Female subject is either not of childbearing potential or is practicing a relevant method of birth control.
* Subject is judged to be in good general health.
* Subjects must be able and willing to provide written informed consent.
* Subjects must be able and willing to self-administer subcutaneous (SC) injections or have a qualified person available to administer SC injections.

Exclusion Criteria:

* Treatment with intra-articular or parenteral administration of corticosteroids in the preceding 4 weeks.
* Oral prednisone or prednisone equivalent > 10 mg/day at baseline.
* Joint surgery within the preceding two months.
* History of acute inflammatory joint disease other than RA.
* Treatment with any investigational drug within 30 days or 5 half lives, whichever is longer prior to study entry.
* Poorly controlled medical condition, which would put the subject at risk by participation in the study.
* History of clinically significant hematologic, renal or liver disease.
* Diagnosis of, or history suggestive of, central nervous system (CNS) demyelinating disease.
* History of cancer or lymphoproliferative disease other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma or localized carcinoma of the cervix.
* History of listeriosis, histoplasmosis, untreated tuberculosis (TB), persistent chronic infections, or recent active infections.
* Known immune deficiency or human immunodeficiency virus (HIV).
* Female who is pregnant or breast-feeding or considering becoming pregnant or breast feeding during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Heimburger, MD, Study Director — AbbVie AB
Locations (8):
- Sweden (8):
  - Site Reference ID/Investigator# 22062, Linköping
  - Site Reference ID/Investigator# 14022, Lund
  - Site Reference ID/Investigator# 14023, Malmo
  - Site Reference ID/Investigator# 14301, Oskarström
  - Site Reference ID/Investigator# 20241, Skövde
  - Site Reference ID/Investigator# 4918, Stockholm
  - Site Reference ID/Investigator# 14021, Stockholm
  - Site Reference ID/Investigator# 14302, Uppsala

REFERENCES:
- [Derived] Chatzidionysiou K, Turesson C, Teleman A, Knight A, Lindqvist E, Larsson P, Coster L, Forslind K, van Vollenhoven R, Heimburger M. A multicentre, randomised, controlled, open-label pilot study on the feasibility of discontinuation of adalimumab in established patients with rheumatoid arthritis in stable clinical remission. RMD Open. 2016 Jan 14;2(1):e000133. doi: 10.1136/rmdopen-2015-000133. eCollection 2016. PMID 26819752
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with rheumatoid arthritis (RA) treated with adalimumab plus methotrexate and in remission for at least the past 3 months were enrolled from 8 investigative sites in Sweden.
Pre-assignment Details: Participants were randomized to continue or discontinue adalimumab treatment for 52 weeks. After the final visit an observational extension period ensued where patients were treated at the discretion of the investigator. The observational extension period lasted until a follow-up visit scheduled at Weeks 104 - 156 (average Week 125).
Period: Randomized Phase
Arm/Group | Adalimumab + MTX | Methotrexate
Started | 17 | 16
Received Rescue Therapy | 0 | 9
Completed | 15 | 11 (Includes participants who received rescue therapy & follow-up for 12 weeks)
Not Completed | 2 | 5
Not completed — Did not meet eligibility criteria | 1 | 0
Not completed — Reduced methotrexate dose | 1 | 2
Not completed — Patient refused rescue therapy | 0 | 3
Period: Observation Phase
Arm/Group | Adalimumab + MTX | Methotrexate
Started | 16 (The observation phase was open to all participants) | 15 (The observation phase was open to all participants)
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab + MTX | Methotrexate | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (13.0) | 61.3 (9.9) | 56.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  Sweden | 17 | 16 | 33
Disease duration [Mean (Standard Deviation); unit: years] | 10.4 (8.9) | 13.2 (12.5) | 11.7 (10.7)
Disease Activity Score (DAS) 28 [Mean (Standard Deviation); unit: units on a scale] — The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity.
  units on a scale | 1.98 (0.48) | 1.73 (0.61) | 1.86 (0.55)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Remission at Week 28
Description: Remission is defined as a Disease Activity Score (DAS)28 of less than 2.6. The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein (CRP), and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity.
  In this analysis participants in the methotrexate treatment group with a DAS28 score ≥ 2.6 (and thus allocated to rescue therapy with adalimumab) prior to Week 28 were considered not to be in remission at Week 28. Also, participants who did not complete 28 weeks were considered not in remission.
Time Frame: Week 28
Population: Full analysis set (FAS), defined as all participants who received at least one dose of adalimumab and/or methotrexate and had at least one post-baseline observation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
percentage of participants | 87.5 [61.7 to 98.4] | 18.8 [4.0 to 45.6]

2. Secondary Outcome: Percentage of Participants in Remission at Week 52
Description: Remission is defined as a Disease Activity Score (DAS)28 of less than 2.6. The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein (CRP), and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity.
  In this analysis participants in the methotrexate treatment group with a DAS28 score ≥ 2.6 (and thus allocated to rescue therapy with adalimumab) prior to Week 52 were considered not to be in remission at Week 52. Also, participants who did not complete 52 weeks were considered not in remission.
Time Frame: Week 52
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
percentage of participants | 81.3 [54.4 to 96.0] | 12.5 [1.6 to 38.3]

3. Secondary Outcome: Percentage of Participants in Remission at Week 52 (FAS2)
Description: Remission is defined as a Disease Activity Score (DAS)28 of less than 2.6. The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein (CRP), and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity. Also, participants who did not complete 52 weeks were considered not in remission.
  In this analysis participants in the methotrexate treatment group with a DAS28 score ≥ 2.6 (and thus allocated to rescue therapy with adalimumab) prior to Week 52 were considered not to be in remission at Week 52.
Time Frame: Week 52
Population: Full analysis set 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 15
percentage of participants | 81.3 [54.4 to 96.0] | 13.3 [1.7 to 40.5]

4. Secondary Outcome: Number of Participants With a Flare
Description: Flare is defined as DAS28 ≥2.6 or an increase from Baseline in the DAS28 of greater than 1.2 units. The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein (CRP), and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity.
Time Frame: Baseline and Weeks 4, 8, 12, 20, 28, 36, 44, and 52
Population: Full analysis set; N indicates the number of participants with available data at each time point.
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Week 4 (N= 16, 14) | 2 | 3
  Week 8 (N= 16, 13) | 0 | 3
  Week 12 (N= 16, 12) | 4 | 4
  Week 20 (N= 16, 8) | 3 | 2
  Week 28 (N=15, 8) | 1 | 3
  Week 36 (N= 15, 5) | 4 | 0
  Week 44 (N=15, 3) | 2 | 0
  Week 52 (N= 15, 2) | 2 | 0

5. Secondary Outcome: Percentage of Participants With Response to Adalimumab Treatment (Return to Baseline DAS28 + ≤ 10%) After a Flare
Description: For participants with a flare and treated with adalimumab rescue therapy, response was defined as return to Baseline DAS28 + ≤ 10% after reinstitution of adalimumab (rescue therapy).
  The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein (CRP), and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity.
Time Frame: 1 to 4 weeks, 5 to 8 weeks, 9 to 12 weeks, and 13 to 16 weeks after reinstitution of adalimumab rescue therapy
Population: Full analysis set participants in the methotrexate treatment group with a flare who were reinstituted adalimumab rescue therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 0 | 9
percentage of participants
  1 - 4 weeks after reinstitution |  | 33.3 [7.5 to 70.1]
  5 - 8 weeks after reinstitution |  | 0 [0.0 to 33.6]
  9 - 12 weeks after reinstitution |  | 22.2 [2.8 to 60.0]
  13 - 16 weeks after reinstitution |  | 11.1 [0.3 to 48.2]

6. Secondary Outcome: Percentage of Participants With Response to Adalimumab Treatment (DAS28 <2.6 or DAS28 Decrease >1.2 Units) After a Flare
Description: For participants with a flare and treated with adalimumab rescue therapy, response was defined as DAS28 less than 2.6 or DAS28 decrease of greater than 1.2 units after reinstitution of adalimumab (rescue therapy). The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein (CRP), and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity.
Time Frame: 1 to 4 weeks, 5 to 8 weeks, 9 to 12 weeks, and 13 to 16 weeks after reinstitution of adalimumab rescue therapy
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 0 | 9
percentage of participants
  1 - 4 weeks after reinstitution |  | 66.7 [29.9 to 92.5]
  5 - 8 weeks after reinstitution |  | 0 [0.0 to 33.6]
  9 - 12 weeks after reinstitution |  | 22.2 [2.8 to 60.0]
  13 - 16 weeks after reinstitution |  | 0 [0.0 to 33.6]

7. Secondary Outcome: Health Assessment Questionnaire (HAQ) Total Score by Visit
Description: Physical function was evaluated using the Health Assessment Questionnaire - Disability Index (HAQ-DI), a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. HAQ remission indicating normal physical function is defined by HAQ-DI < 0.5.
Time Frame: Baseline and Weeks 4, 8, 12, 20, 28, 36, 44, 52, and 104-156 (extension period visit)
Population: Full analysis set; N indicates the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
units on a scale
  Baseline (N=16, 16) | 0.35 (0.40) | 0.39 (0.26)
  Week 4 (N= 16, 15) | 0.35 (0.41) | 0.42 (0.37)
  Week 8 (N=16, 15) | 0.34 (0.39) | 0.39 (0.31)
  Week 12 (N=16, 13) | 0.31 (0.40) | 0.50 (0.37)
  Week 20 (N=16, 10) | 0.37 (0.42) | 0.54 (0.41)
  Week 28 (N=16, 8) | 0.36 (0.41) | 0.41 (0.36)
  Week 36 (N=15, 5) | 0.37 (0.44) | 0.45 (0.27)
  Week 44 (N=15, 5) | 0.38 (0.43) | 0.48 (0.29)
  Week 52 (N=15, 2) | 0.44 (0.43) | 0.50 (0.00)
  Weeks 104-156 (N=16, 15) | 0.39 (0.47) | 0.42 (0.33)

8. Secondary Outcome: European Quality of Life-5 Dimensions (EQ-5D) Mobility Score by Visit
Description: The EQ-5D is an international, standardized, generic instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their mobility health state:
  Level 1: I have no problems in walking about;
  Level 2: I have some problems in walking about;
  Level 3: I am confined to bed.
Time Frame: Baseline and Weeks 4, 8, 12, 20, 28, 36, 44, 52, and 104-156 (extension period visit)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Level 1 | 12 | 13
  Baseline: Level 2 | 4 | 2
  Baseline: Level 3 | 0 | 0
  Baseline: Missing | 0 | 1
  Week 4: Level 1 | 13 | 11
  Week 4: Level 2 | 3 | 3
  Week 4: Level 3 | 0 | 0
  Week 4: Missing | 0 | 2
  Week 8: Level 1 | 11 | 10
  Week 8: Level 2 | 5 | 3
  Week 8: Level 3 | 0 | 0
  Week 8: Missing | 0 | 3
  Week 12: Level 1 | 13 | 10
  Week 12: Level 2 | 3 | 2
  Week 12: Level 3 | 0 | 0
  Week 12: Missing | 0 | 4
  Week 20: Level 1 | 12 | 6
  Week 20: Level 2 | 4 | 2
  Week 20: Level 3 | 0 | 0
  Week 20: Missing | 0 | 8
  Week 28: Level 1 | 10 | 7
  Week 28: Level 2 | 5 | 1
  Week 28: Level 3 | 0 | 0
  Week 28: Missing | 1 | 8
  Week 36: Level 1 | 10 | 5
  Week 36: Level 2 | 5 | 0
  Week 36: Level 3 | 0 | 0
  Week 36: Missing | 1 | 11
  Week 44: Level 1 | 11 | 3
  Week 44: Level 2 | 4 | 0
  Week 44: Level 3 | 0 | 0
  Week 44: Missing | 1 | 13
  Week 52: Level 1 | 10 | 2
  Week 52: Level 2 | 5 | 0
  Week 52: Level 3 | 0 | 0
  Week 52: Missing | 1 | 14
  Weeks 104-156: Level 1 | 10 | 13
  Weeks 104-156: Level 2 | 6 | 1
  Weeks 104-156: Level 3 | 0 | 0
  Weeks 104-156: Missing | 0 | 2

9. Secondary Outcome: European Quality of Life-5 Dimensions (EQ-5D) Self-care Score by Visit
Description: The EQ-5D is an international, standardized, generic instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their self-care health state:
  Level 1: I have no problems with self-care;
  Level 2: I have some problems washing or dressing myself;
  Level 3: I am unable to wash or dress myself.
Time Frame: Baseline and Weeks 4, 8, 12, 20, 28, 36, 44, 52, and 104-156 (extension period visit)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Level 1 | 15 | 16
  Baseline: Level 2 | 1 | 0
  Baseline: Level 3 | 0 | 0
  Baseline: Missing | 0 | 0
  Week 4: Level 1 | 16 | 12
  Week 4: Level 2 | 0 | 1
  Week 4: Level 3 | 0 | 1
  Week 4: Missing | 0 | 2
  Week 8: Level 1 | 16 | 13
  Week 8: Level 2 | 0 | 0
  Week 8: Level 3 | 0 | 0
  Week 8: Missing | 0 | 3
  Week 12: Level 1 | 15 | 9
  Week 12: Level 2 | 1 | 2
  Week 12: Level 3 | 0 | 1
  Week 12: Missing | 0 | 4
  Week 20: Level 1 | 16 | 8
  Week 20: Level 2 | 0 | 0
  Week 20: Level 3 | 0 | 0
  Week 20: Missing | 0 | 8
  Week 28: Level 1 | 14 | 8
  Week 28: Level 2 | 1 | 0
  Week 28: Level 3 | 0 | 0
  Week 28: Missing | 1 | 8
  Week 36: Level 1 | 15 | 5
  Week 36: Level 2 | 0 | 0
  Week 36: Level 3 | 0 | 0
  Week 36: Missing | 1 | 11
  Week 44: Level 1 | 14 | 2
  Week 44: Level 2 | 1 | 1
  Week 44: Level 3 | 0 | 0
  Week 44: Missing | 1 | 13
  Week 52: Level 1 | 15 | 2
  Week 52: Level 2 | 0 | 0
  Week 52: Level 3 | 0 | 0
  Week 52: Missing | 1 | 14
  Weeks 104-156: Level 1 | 16 | 14
  Weeks 104-156: Level 2 | 0 | 0
  Weeks 104-156: Level 3 | 0 | 0
  Weeks 104-156: Missing | 0 | 2

10. Primary Outcome: Percentage of Participants in Remission at Week 28 in the Full Analysis Set 2 (FAS2)
Description: as for outcome 1
Time Frame: Week 28
Population: Full analysis set 2 (FAS2), defined as participants in the full analysis set who completed at least 28 weeks of the study or completed the study until flare, whichever occurs first.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 15
percentage of participants | 87.5 [61.7 to 98.4] | 20.0 [4.3 to 48.1]

11. Secondary Outcome: European Quality of Life-5 Dimensions (EQ-5D) Usual Activities Score by Visit
Description: The EQ-5D is an international, standardized, generic instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their health state with regard to usual activities (work, study, housework, family, or leisure activities):
  Level 1: I have no problems performing my usual activities;
  Level 2: I have some problems performing my usual activities;
  Level 3: I am unable to perform my usual activities.
Time Frame: Baseline and Weeks 4, 8, 12, 20, 28, 36, 44, 52, and 104-156 (extension period visit)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Level 1 | 14 | 15
  Baseline: Level 2 | 2 | 1
  Baseline: Level 3 | 0 | 0
  Baseline: Missing | 0 | 0
  Week 4: Level 1 | 14 | 13
  Week 4: Level 2 | 2 | 1
  Week 4: Level 3 | 0 | 0
  Week 4: Missing | 0 | 2
  Week 8: Level 1 | 15 | 12
  Week 8: Level 2 | 1 | 1
  Week 8: Level 3 | 0 | 0
  Week 8: Missing | 0 | 3
  Week 12: Level 1 | 14 | 9
  Week 12: Level 2 | 2 | 3
  Week 12: Level 3 | 0 | 0
  Week 12: Missing | 0 | 4
  Week 20: Level 1 | 13 | 7
  Week 20: Level 2 | 3 | 1
  Week 20: Level 3 | 0 | 0
  Week 20: Missing | 0 | 8
  Week 28: Level 1 | 13 | 7
  Week 28: Level 2 | 2 | 1
  Week 28: Level 3 | 0 | 0
  Week 28: Missing | 1 | 8
  Week 36: Level 1 | 12 | 5
  Week 36: Level 2 | 3 | 0
  Week 36: Level 3 | 0 | 0
  Week 36: Missing | 1 | 11
  Week 44: Level 1 | 12 | 2
  Week 44: Level 2 | 3 | 1
  Week 44: Level 3 | 0 | 0
  Week 44: Missing | 1 | 13
  Week 52: Level 1 | 12 | 1
  Week 52: Level 2 | 3 | 1
  Week 52: Level 3 | 0 | 0
  Week 52: Missing | 1 | 14
  Weeks 104-156: Level 1 | 13 | 14
  Weeks 104-156: Level 2 | 3 | 0
  Weeks 104-156: Level 3 | 0 | 0
  Weeks 104-156: Missing | 0 | 2

12. Secondary Outcome: European Quality of Life-5 Dimensions (EQ-5D) Pain/Discomfort Score by Visit
Description: The EQ-5D is an international, standardized, generic instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their pain/discomfort health state:
  Level 1: I have no pain or discomfort;
  Level 2: I have moderate pain or discomfort;
  Level 3: I have extreme pain or discomfort.
Time Frame: Baseline and Weeks 4, 8, 12, 20, 28, 36, 44, 52, and 104-156 (extension period visit)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Level 1 | 6 | 3
  Baseline: Level 2 | 10 | 13
  Baseline: Level 3 | 0 | 0
  Baseline: Missing | 0 | 0
  Week 4: Level 1 | 8 | 2
  Week 4: Level 2 | 8 | 12
  Week 4: Level 3 | 0 | 0
  Week 4: Missing | 0 | 2
  Week 8: Level 1 | 7 | 1
  Week 8: Level 2 | 9 | 12
  Week 8: Level 3 | 0 | 0
  Week 8: Missing | 0 | 3
  Week 12: Level 1 | 8 | 0
  Week 12: Level 2 | 8 | 12
  Week 12: Level 3 | 0 | 0
  Week 12: Missing | 0 | 4
  Week 20: Level 1 | 7 | 0
  Week 20: Level 2 | 9 | 8
  Week 20: Level 3 | 0 | 0
  Week 20: Missing | 0 | 8
  Week 28: Level 1 | 5 | 3
  Week 28: Level 2 | 10 | 5
  Week 28: Level 3 | 0 | 0
  Week 28: Missing | 1 | 8
  Week 36: Level 1 | 8 | 1
  Week 36: Level 2 | 7 | 4
  Week 36: Level 3 | 0 | 0
  Week 36: Missing | 1 | 11
  Week 44: Level 1 | 7 | 0
  Week 44: Level 2 | 8 | 3
  Week 44: Level 3 | 0 | 0
  Week 44: Missing | 1 | 13
  Week 52: Level 1 | 5 | 0
  Week 52: Level 2 | 10 | 2
  Week 52: Level 3 | 0 | 0
  Week 52: Missing | 1 | 14
  Weeks 104-156: Level 1 | 8 | 3
  Weeks 104-156: Level 2 | 8 | 11
  Weeks 104-156: Level 3 | 0 | 0
  Weeks 104-156: Missing | 0 | 2

13. Secondary Outcome: European Quality of Life-5 Dimensions (EQ-5D) Anxiety/Depression Score by Visit
Description: The EQ-5D is an international, standardized, generic instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their anxiety/depression health state:
  Level 1: I am not anxious or depressed;
  Level 2: I am moderately anxious or depressed;
  Level 3: I am extremely anxious or depressed.
Time Frame: Baseline and Weeks 4, 8, 12, 20, 28, 36, 44, 52, and 104-156 (extension period visit)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Level 1 | 14 | 12
  Baseline: Level 2 | 2 | 4
  Baseline: Level 3 | 0 | 0
  Baseline: Missing | 0 | 0
  Week 4: Level 1 | 13 | 10
  Week 4: Level 2 | 3 | 4
  Week 4: Level 3 | 0 | 0
  Week 4: Missing | 0 | 2
  Week 8: Level 1 | 13 | 11
  Week 8: Level 2 | 3 | 2
  Week 8: Level 3 | 0 | 0
  Week 8: Missing | 0 | 3
  Week 12: Level 1 | 14 | 8
  Week 12: Level 2 | 2 | 4
  Week 12: Level 3 | 0 | 0
  Week 12: Missing | 0 | 4
  Week 20: Level 1 | 13 | 6
  Week 20: Level 2 | 3 | 2
  Week 20: Level 3 | 0 | 0
  Week 20: Missing | 0 | 8
  Week 28: Level 1 | 13 | 6
  Week 28: Level 2 | 2 | 2
  Week 28: Level 3 | 0 | 0
  Week 28: Missing | 1 | 8
  Week 36: Level 1 | 12 | 4
  Week 36: Level 2 | 3 | 1
  Week 36: Level 3 | 0 | 0
  Week 36: Missing | 1 | 11
  Week 44: Level 1 | 13 | 2
  Week 44: Level 2 | 2 | 1
  Week 44: Level 3 | 0 | 0
  Week 44: Missing | 1 | 13
  Week 52: Level 1 | 11 | 1
  Week 52: Level 2 | 4 | 1
  Week 52: Level 3 | 0 | 0
  Week 52: Missing | 1 | 14
  Weeks 104-156: Level 1 | 11 | 13
  Weeks 104-156: Level 2 | 5 | 1
  Weeks 104-156: Level 3 | 0 | 0
  Weeks 104-156: Missing | 0 | 2

14. Secondary Outcome: European Quality of Life-5 Dimensions (EQ-5D) Visual Analog Scale (VAS) by Visit
Description: The EQ-5D is an international, standardized, generic instrument for describing and evaluating health status. Health status is assessed by patients evaluating their health on a vertical, visual analog scale from 0 to 100 where the endpoints are labeled 'Worst imaginable health state' (0) and 'Best imaginable health state' (100).
Time Frame: Baseline and Weeks 4, 8, 12, 20, 28, 36, 44, 52, and 104-156 (extension period visit)
Population: Full analysis set; N indicates the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
units on a scale
  Baseline (N=16, 16) | 88.2 (9.3) | 89.9 (7.5)
  Week 4 (N= 16, 14) | 85.6 (13.4) | 83.2 (19.1)
  Week 8 (N=16, 13) | 88.4 (11.1) | 82.8 (20.7)
  Week 12 (N=16, 12) | 89.9 (12.4) | 82.9 (11.6)
  Week 20 (N=16, 8) | 87.1 (14.9) | 90.4 (6.0)
  Week 28 (N=15, 8) | 88.0 (10.3) | 90.8 (7.2)
  Week 36 (N=15, 5) | 80.5 (22.8) | 90.6 (6.3)
  Week 44 (N=15, 3) | 85.9 (12.2) | 88.7 (9.0)
  Week 52 (N=15, 2) | 86.2 (13.0) | 89.0 (12.7)
  Weeks 104-156 (N=16, 15) | 85.6 (15.0) | 86.0 (13.7)

15. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Scale by Visit
Description: The FACIT-Fatigue questionnaire is a self-administered patient questionnaire that consists of 13 questions designed to measure the degree of fatigue experienced by participants in the previous 7 days. Participants respond to the questions on a scale from 'not at all' (0) to 'very much' (4). The scale score is computed by summing the item scores, after reversing those items that are worded in the negative direction. The FACIT-Fatigue subscale score ranges from 0 to 52, where higher scores represent less fatigue.
Time Frame: Baseline and Weeks 4, 8, 12, 20, 28, 36, 44, 52, and 104-156 (extension period visit)
Population: Full analysis set; N indicates the number of participants with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
units on a scale
  Baseline (N=16, 16) | 45.2 (8.7) | 42.5 (5.0)
  Week 4 (N=16, 14) | 45.3 (6.3) | 43.6 (6.3)
  Week 8 (N=15, 13) | 46.9 (5.9) | 44.9 (4.8)
  Week 12 (N=16, 12) | 47.4 (4.9) | 41.7 (6.9)
  Week 20 (N=16, 8) | 46.7 (5.7) | 43.2 (6.5)
  Week 28 (N=15, 8) | 46.1 (7.4) | 42.9 (8.9)
  Week 36 (N=15, 5) | 45.4 (8.4) | 43.8 (10.1)
  Week 44 (N=15, 3) | 46.6 (6.7) | 41.3 (16.8)
  Week 52 (N=15, 2) | 45.7 (8.4) | 37.5 (17.7)
  Weeks 104-156 (N=16, 15) | 45.9 (6.8) | 45.3 (6.0)

16. Secondary Outcome: Work Instability Score (WIS) for RA: I'm Getting up Earlier Because of Arthritis
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 1, participants selected either Yes or No if the following statement currently applied to them or not: I'm getting up earlier because of the arthritis.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 2 | 1
  Baseline: No | 10 | 7
  Baseline: Missing | 4 | 8
  Week 12: Yes | 1 | 0
  Week 12: No | 10 | 7
  Week 12: Missing | 5 | 9
  Week 28: Yes | 2 | 0
  Week 28: No | 10 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 3 | 0
  Week 52: No | 10 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 0 | 0
  Weeks 104-156: No | 12 | 6
  Weeks 104-156: Missing | 4 | 10

17. Secondary Outcome: Work Instability Score (WIS) for RA: I Get Very Stiff at Work
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 2, participants selected either Yes or No if the following statement currently applied to them or not: I get very stiff at work.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 1 | 0
  Baseline: No | 11 | 7
  Baseline: Missing | 4 | 9
  Week 12: Yes | 1 | 1
  Week 12: No | 10 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 1 | 0
  Week 28: No | 11 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 1 | 1
  Week 52: No | 12 | 0
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 1 | 1
  Weeks 104-156: No | 11 | 5
  Weeks 104-156: Missing | 4 | 10

18. Secondary Outcome: Work Instability Score (WIS) for RA: I'm Finding my Job is About All I Can Manage
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 3, participants selected either Yes or No if the following statement currently applied to them or not: I'm finding my job is about all I can manage.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 2 | 1
  Baseline: No | 10 | 6
  Baseline: Missing | 4 | 9
  Week 12: Yes | 2 | 1
  Week 12: No | 9 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 2 | 2
  Week 28: No | 10 | 1
  Week 28: Missing | 4 | 13
  Week 52: Yes | 2 | 1
  Week 52: No | 11 | 0
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 3 | 1
  Weeks 104-156: No | 9 | 5
  Weeks 104-156: Missing | 4 | 10

19. Secondary Outcome: Work Instability Score (WIS) for RA: The Stress of my Job Makes my Arthritis Flare
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 4, participants selected either Yes or No if the following statement currently applied to them or not: The stress of my job makes my arthritis flare.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 3 | 0
  Baseline: No | 9 | 7
  Baseline: Missing | 4 | 9
  Week 12: Yes | 2 | 1
  Week 12: No | 9 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 1 | 0
  Week 28: No | 11 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 2 | 0
  Week 52: No | 11 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 1 | 0
  Weeks 104-156: No | 11 | 6
  Weeks 104-156: Missing | 4 | 10

20. Secondary Outcome: Work Instability Score (WIS) for RA: I'm Finding Any Pressure on my Hands is a Problem
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 5, participants selected either Yes or No if the following statement currently applied to them or not: I'm finding any pressure on my hands is a problem.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 2 | 1
  Baseline: No | 10 | 6
  Baseline: Missing | 4 | 9
  Week 12: Yes | 2 | 1
  Week 12: No | 9 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 3 | 1
  Week 28: No | 9 | 2
  Week 28: Missing | 4 | 13
  Week 52: Yes | 3 | 1
  Week 52: No | 10 | 0
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 2 | 1
  Weeks 104-156: No | 10 | 5
  Weeks 104-156: Missing | 4 | 10

21. Secondary Outcome: Work Instability Score (WIS) for RA: I Get Good Days and Bad Days at Work
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 6, participants selected either Yes or No if the following statement currently applied to them or not: I get good days and bad days at work.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 6 | 4
  Baseline: No | 6 | 3
  Baseline: Missing | 4 | 9
  Week 12: Yes | 5 | 2
  Week 12: No | 6 | 2
  Week 12: Missing | 5 | 12
  Week 28: Yes | 6 | 1
  Week 28: No | 6 | 2
  Week 28: Missing | 4 | 13
  Week 52: Yes | 9 | 1
  Week 52: No | 4 | 0
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 5 | 3
  Weeks 104-156: No | 7 | 3
  Weeks 104-156: Missing | 4 | 10

22. Secondary Outcome: Work Instability Score (WIS) for RA: I Can Get my Job Done, I'm Just a Lot Slower
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 7, participants selected either Yes or No if the following statement currently applied to them or not: I can get my job done, I'm just a lot slower.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 3 | 1
  Baseline: No | 9 | 6
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 2 | 1
  Week 28: No | 10 | 2
  Week 28: Missing | 4 | 13
  Week 52: Yes | 3 | 0
  Week 52: No | 10 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 3 | 1
  Weeks 104-156: No | 9 | 5
  Weeks 104-156: Missing | 4 | 10

23. Secondary Outcome: Work Instability Score (WIS) for RA: If I Don't Reduce my Hours I May Have to Give up Work
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 8, participants selected either Yes or No if the following statement currently applied to them or not: If I don't reduce my hours I may have to give up work.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 3 | 1
  Baseline: No | 9 | 6
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 2 | 0
  Week 28: No | 10 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 3 | 0
  Week 52: No | 10 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 2 | 1
  Weeks 104-156: No | 10 | 5
  Weeks 104-156: Missing | 4 | 10

24. Secondary Outcome: Work Instability Score (WIS) for RA: I am Very Worried About my Ability to Keep Working
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 9, participants selected either Yes or No if the following statement currently applies to them or not: I am very worried about my ability to keep working.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 2 | 1
  Baseline: No | 10 | 6
  Baseline: Missing | 4 | 9
  Week 12: Yes | 2 | 1
  Week 12: No | 9 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 3 | 0
  Week 28: No | 9 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 1 | 1
  Week 52: No | 12 | 0
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 2 | 1
  Weeks 104-156: No | 10 | 5
  Weeks 104-156: Missing | 4 | 10

25. Secondary Outcome: Work Instability Score (WIS) for RA: I Have Pain or Stiffness All the Time at Work
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 10, participants selected either Yes or No if the following statement currently applies to them or not: I have pain or stiffness all the time at work.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 0 | 0
  Baseline: No | 12 | 7
  Baseline: Missing | 4 | 9
  Week 12: Yes | 0 | 0
  Week 12: No | 11 | 4
  Week 12: Missing | 5 | 12
  Week 28: Yes | 0 | 0
  Week 28: No | 12 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 1 | 0
  Week 52: No | 12 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 1 | 0
  Weeks 104-156: No | 11 | 6
  Weeks 104-156: Missing | 4 | 10

26. Secondary Outcome: Work Instability Score (WIS) for RA: I Don't Have the Stamina to Work Like I Used to
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 11, participants selected either Yes or No if the following statement currently applies to them or not: I don't have the stamina to work like I used to.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 5 | 2
  Baseline: No | 7 | 5
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 4 | 0
  Week 28: No | 8 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 5 | 0
  Week 52: No | 8 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 4 | 4
  Weeks 104-156: No | 8 | 2
  Weeks 104-156: Missing | 4 | 10

27. Secondary Outcome: Work Instability Score (WIS) for RA: I Have Used my Vacation so That I Don't Have to Take Sick Leave
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 12, participants selected either Yes or No if the following statement currently applies to them or not: I have used my vacation so that I don't have to take sick leave.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 5 | 2
  Baseline: No | 7 | 5
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 4 | 0
  Week 28: No | 8 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 5 | 0
  Week 52: No | 8 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 4 | 4
  Weeks 104-156: No | 8 | 2
  Weeks 104-156: Missing | 4 | 10

28. Secondary Outcome: Work Instability Score (WIS) for RA: I Push Myself to go to Work Because I Don't Want to Give in to the Arthritis
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 13, participants selected either Yes or No if the following statement currently applies to them or not: I push myself to go to work because I don't want to give in to the arthritis.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 5 | 2
  Baseline: No | 7 | 5
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 4 | 0
  Week 28: No | 8 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 5 | 0
  Week 52: No | 8 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 4 | 4
  Weeks 104-156: No | 8 | 2
  Weeks 104-156: Missing | 4 | 10

29. Secondary Outcome: Work Instability Score (WIS) for RA: Sometimes I Can't Face Being at Work All Day
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 14, participants selected either Yes or No if the following statement currently applies to them or not: Sometimes I can't face being at work all day.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 5 | 2
  Baseline: No | 7 | 5
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 4 | 0
  Week 28: No | 8 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 5 | 0
  Week 52: No | 8 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 4 | 4
  Weeks 104-156: No | 8 | 2
  Weeks 104-156: Missing | 4 | 10

30. Secondary Outcome: Work Instability Score (WIS) for RA: I Have to Say No to Certain Things at Work
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 15, participants selected either Yes or No if the following statement currently applies to them or not: I have to say no to certain things at work.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 5 | 2
  Baseline: No | 7 | 5
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 4 | 0
  Week 28: No | 8 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 5 | 0
  Week 52: No | 8 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 4 | 4
  Weeks 104-156: No | 8 | 2
  Weeks 104-156: Missing | 4 | 10

31. Secondary Outcome: Work Instability Score (WIS) for RA: I've Got to Watch How Much I do Certain Things at Work
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 16, participants selected either Yes or No if the following statement currently applies to them or not: I've got to watch how much I do certain things at work.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 5 | 2
  Baseline: No | 7 | 5
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 4 | 0
  Week 28: No | 8 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 5 | 0
  Week 52: No | 8 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 4 | 4
  Weeks 104-156: No | 8 | 2
  Weeks 104-156: Missing | 4 | 10

32. Secondary Outcome: Work Instability Score (WIS) for RA: I Have Great Difficulty Opening Some of the Doors at Work
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 17, participants selected either Yes or No if the following statement currently applies to them or not: I have great difficulty opening some of the doors at work.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 5 | 2
  Baseline: No | 7 | 5
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 4 | 0
  Week 28: No | 8 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 5 | 0
  Week 52: No | 8 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 4 | 4
  Weeks 104-156: No | 8 | 2
  Weeks 104-156: Missing | 4 | 10

33. Secondary Outcome: Work Instability Score (WIS) for RA: I Have to Allow Myself Extra Time to do Some Jobs
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 18, participants selected either Yes or No if the following statement currently applies to them or not: I have to allow myself extra time to do some jobs.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 5 | 2
  Baseline: No | 7 | 5
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 4 | 0
  Week 28: No | 8 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 5 | 0
  Week 52: No | 8 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 4 | 4
  Weeks 104-156: No | 8 | 2
  Weeks 104-156: Missing | 4 | 10

34. Secondary Outcome: Work Instability Score (WIS) for RA: It's Very Frustrating Because I Can't Always do Things at Work
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 19, participants selected either Yes or No if the following statement currently applies to them or not: It's very frustrating because I can't always do things at work.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 5 | 2
  Baseline: No | 7 | 5
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 4 | 0
  Week 28: No | 8 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 5 | 0
  Week 52: No | 8 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 4 | 4
  Weeks 104-156: No | 8 | 2
  Weeks 104-156: Missing | 4 | 10

35. Secondary Outcome: Work Instability Score (WIS) for RA: I Feel I May Have to Give up Work
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 20, participants selected either Yes or No if the following statement currently applies to them or not: I feel I may have to give up work.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 5 | 2
  Baseline: No | 7 | 5
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 4 | 0
  Week 28: No | 8 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 5 | 0
  Week 52: No | 8 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 4 | 4
  Weeks 104-156: No | 8 | 2
  Weeks 104-156: Missing | 4 | 10

36. Secondary Outcome: Work Instability Score (WIS) for RA: I Get on With the Work But Afterwards I Have a Lot of Pain
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 21, participants selected either Yes or No if the following statement currently applies to them or not: I get on with the work but afterwards I have a lot of pain.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 5 | 2
  Baseline: No | 7 | 5
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 4 | 0
  Week 28: No | 8 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 5 | 0
  Week 52: No | 8 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 4 | 4
  Weeks 104-156: No | 8 | 2
  Weeks 104-156: Missing | 4 | 10

37. Secondary Outcome: Work Instability Score (WIS) for RA: When I'm Feeling Tired All the Time Work is a Grind
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 22, participants selected either Yes or No if the following statement currently applies to them or not: When I'm feeling tired all the time work is a grind.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 5 | 2
  Baseline: No | 7 | 5
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 4 | 0
  Week 28: No | 8 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 5 | 0
  Week 52: No | 8 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 4 | 4
  Weeks 104-156: No | 8 | 2
  Weeks 104-156: Missing | 4 | 10

38. Secondary Outcome: Work Instability Score (WIS) for RA: I'd Like Another Job But I am Restricted to What I Can do
Description: Work Instability (defined as the mismatch between the person's abilities and the demands of work) Score is a 23-item questionnaire designed to indicate the participant's level of risk for work disability. In question 23, participants selected either Yes or No if the following statement currently applied to them or not: I'd like another job but I am restricted to what I can do.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 5 | 2
  Baseline: No | 7 | 5
  Baseline: Missing | 4 | 9
  Week 12: Yes | 4 | 1
  Week 12: No | 7 | 3
  Week 12: Missing | 5 | 12
  Week 28: Yes | 4 | 0
  Week 28: No | 8 | 3
  Week 28: Missing | 4 | 13
  Week 52: Yes | 5 | 0
  Week 52: No | 8 | 1
  Week 52: Missing | 3 | 15
  Weeks 104-156: Yes | 4 | 4
  Weeks 104-156: No | 8 | 2
  Weeks 104-156: Missing | 4 | 10

39. Secondary Outcome: Work Productivity and Activity Impairment (WPAI): Currently Employed
Description: The Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) questionnaire was used to assess work and activity impairment due to symptoms of rheumatoid arthritis in the last 7 days. The self-administered questionnaire consists of 6 questions. Question 1 asks participants to indicate if they are currently employed or working for pay (Yes or No).
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
participants
  Baseline: Yes | 10 | 7
  Baseline: No | 5 | 8
  Baseline: Missing | 1 | 1
  Week 12: Yes | 9 | 4
  Week 12: No | 6 | 8
  Week 12: Missing | 1 | 4
  Week 28: Yes | 10 | 3
  Week 28: No | 5 | 5
  Week 28: Missing | 1 | 8
  Week 52: Yes | 12 | 1
  Week 52: No | 3 | 1
  Week 52: Missing | 1 | 14
  Weeks 104-156: Yes | 9 | 5
  Weeks 104-156: No | 5 | 10
  Weeks 104-156: Missing | 2 | 1

40. Secondary Outcome: Work Productivity and Activity Impairment (WPAI): Hours Missed From Work
Description: The Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) questionnaire was used to assess work and activity impairment due to symptoms of rheumatoid arthritis in the last 7 days. The self-administered questionnaire consists of 6 questions. Question 2 asks participants who are employed or working for pay to indicate the number of hours missed from work due to problems associated with their rheumatoid arthritis.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set participants employed or working for pay; N indicates the number of participants employed or working for pay and with available data at each time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
hours
  Baseline (N=9, 7) | 1.1 (3.3) | 1.1 (3.0)
  Week 12 (N=7, 4) | 1.4 (3.8) | 0.0 (0.0)
  Week 28 (N=10, 3) | 1.4 (3.3) | 6.0 (5.3)
  Week 52 (N=12, 1) | 1.2 (3.0) | 0.0 (NA) — Cannot be calculated due to sample size=1.
  Weeks 104-156 (N=7, 5) | 0.0 (0.0) | 0.0 (0.0)

41. Secondary Outcome: Work Productivity and Activity Impairment (WPAI): Hours Missed From Work for Other Reasons
Description: The Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) questionnaire was used to assess work and activity impairment due to symptoms of rheumatoid arthritis in the last 7 days. The self-administered questionnaire consists of 6 questions. Question 3 asks participants who are employed or working for pay to indicate the number of hours missed from work due to reasons other than rheumatoid arthritis.
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
hours
  Baseline (N=8, 7) | 3.8 (9.1) | 5.0 (8.9)
  Week 12 (N=8, 4) | 11.9 (16.0) | 8.3 (13.4)
  Week 28 (N=10, 3) | 3.2 (5.9) | 3.8 (4.0)
  Week 52 (N=12, 1) | 6.3 (11.7) | 16.5 (NA) — Cannot be calculated due to a sample size of 1.
  Weeks 104-156 (N=7, 5) | 2.9 (5.9) | 26.2 (56.9)

42. Secondary Outcome: Work Productivity and Activity Impairment (WPAI): Hours Worked
Description: The Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) questionnaire was used to assess work and activity impairment due to symptoms of rheumatoid arthritis in the last 7 days. The self-administered questionnaire consists of 6 questions. Question 4 asks participants who are employed or working for pay to indicate the number of hours actually worked during the past 7 days.
Time Frame: Baseline and at Weeks 12, 28, 52 and 104-156
Population: Full analysis set participants employed or working for pay and with available data at each time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
hours
  Baseline (N=10, 7) | 31.5 (11.8) | 31.1 (9.7)
  Week 12 (N=6, 3) | 29.8 (11.1) | 38.3 (2.9)
  Week 28 (N=10, 3) | 34.7 (16.4) | 32.7 (9.5)
  Week 52 (N=12, 1) | 30.7 (11.4) | 40.0 (NA) — Cannot be calculated due to a sample size of 1.
  Weeks 104-156 (N=8, 4) | 32.8 (12.8) | 40.3 (16.2)

43. Secondary Outcome: Work Productivity and Activity Impairment (WPAI): Work Productivity
Description: The Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) questionnaire was used to assess work and activity impairment due to symptoms of rheumatoid arthritis in the last 7 days. The self-administered questionnaire consists of 6 questions. Question 5 asks participants who are employed or working for pay to indicate how much their rheumatoid arthritis impaired their productivity while working in the past 7 days on a scale from 0 (no effect) to 10 (completely prevented from working).
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
units on a scale
  Baseline (N=10, 7) | 0.8 (1.9) | 2.1 (2.9)
  Week 12 (N=6, 3) | 1.3 (2.4) | 1.3 (1.5)
  Week 28 (N=10, 3) | 1.0 (1.5) | 1.0 (0.0)
  Week 52 (N=12, 1) | 1.1 (1.8) | 1.0 (NA) — Could not be calculated due to a sample size of 1.
  Weeks 104-156 (N=8, 4) | 1.8 (2.5) | 0.5 (0.6)

44. Secondary Outcome: Work Productivity and Activity Impairment (WPAI): Daily Activities
Description: The Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) questionnaire was used to assess work and activity impairment due to symptoms of rheumatoid arthritis in the last 7 days. The self-administered questionnaire consists of 6 questions. Question 6 asks participants to indicate how much their rheumatoid arthritis affected their ability to do their regular daily activities such as housework, childcare, exercising, shopping, studying, etc, in the past 7 days on a scale from 0 (no effect) to 10 (completely prevented from doing daily activities).
Time Frame: Baseline and at Weeks 12, 28, 52, and 104-156
Population: Full analysis set; N indicates the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
units on a scale
  Baseline (N=14, 15) | 1.6 (1.8) | 1.5 (1.5)
  Week 12 (N=15, 12) | 1.5 (1.7) | 1.8 (1.4)
  Week 28 (N=15, 7) | 1.9 (2.3) | 1.6 (1.3)
  Week 52 (N=15, 2) | 1.7 (1.8) | 1.0 (1.4)
  Weeks 104-156 (N=14, 15) | 2.6 (2.3) | 1.2 (1.0)

45. Secondary Outcome: Change From Baseline in Radiological Modified Total Sharp Score
Description: The van der Heijde modified Total Sharp Score (mTSS) is a measure of the level of joint damage. X-rays of hands and feet were taken at Baseline, Week 52 and the Week 104-156 visit. Joints were scored for erosions on a scale of 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale of 0 (no damage) to 4 (ankylosis or complete dislocation). Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). An increase in mTSS from Baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Baseline, Week 52, and Weeks 104-156
Population: Full analysis set; N indicates the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab + MTX | Methotrexate
Number analyzed (Participants) | 16 | 16
units on a scale
  Change at Week 52 (N=16, 11) | 0.1 (9.4) | -0.8 (13.5)
  Change at Week 104-156 (N=16, 13) | -2.4 (20.9) | -7.2 (15.7)

ADVERSE EVENTS:
Time Frame: From randomization through the observational extension visit (up to Week 156).
Groups:
- Methotrexate-Excluding Rescue: Participants received methotrexate (at least 10 mg/week orally or subcutaneously) alone for 52 weeks and were not reinstituted to adalimumab as rescue treatment. After Week 52 an observational extension period ensued where participants were treated at the discretion of the investigator.
- Methotrexate-Rescue Arm: Participants received methotrexate alone for 52 weeks, but due to an increase in disease activity were reinstituted with adalimumab 40 mg subcutaneously every other week during the 52-week randomized period. After Week 52 an observational extension period ensued where participants were treated at the discretion of the investigator.
- Methotrexate-Including Rescue: Participants received methotrexate (at least 10 mg/week orally or subcutaneously) alone for 52 weeks. Participants with a significant increase in RA disease activity were re-instituted to adalimumab 40 mg every other week (rescue arm). After Week 52 an observational extension period ensued where participants were treated at the discretion of the investigator.
Arm/Group | Adalimumab + MTX | Methotrexate-Excluding Rescue | Methotrexate-Rescue Arm | Methotrexate-Including Rescue
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/7 | 3/9 | 3/16
Other Adverse Events (participants affected / at risk) | 15/17 | 7/7 | 8/9 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab + MTX (N=17) | Methotrexate-Excluding Rescue (N=7) | Methotrexate-Rescue Arm (N=9) | Methotrexate-Including Rescue (N=16)
Chest pain (General disorders) | 0 | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab + MTX (N=17) | Methotrexate-Excluding Rescue (N=7) | Methotrexate-Rescue Arm (N=9) | Methotrexate-Including Rescue (N=16)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Fatigue (General disorders) | 1 | 1 | 1 | 2
Malaise (General disorders) | 1 | 0 | 0 | 0
Nodule (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 4 | 5 | 9
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Shigella infection (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Tooth infection (Infections and infestations) | 2 | 0 | 0 | 0
Upper respiratory tract (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Tooth injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1
Blood thyroid stimulating hormone abnormal (Investigations) | 1 | 0 | 0 | 0
Lipids increased (Investigations) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 1
Urge incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 2
Peripheral coldness (Vascular disorders) | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.